CLINICAL TRIAL: NCT03761875
Title: NK Cell Deregulation in HBV Patients
Acronym: LiNKeB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 87RI18-0021
Record Dates: First submitted 2018-11-12; First posted 2018-12-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis B Virus
Keywords: Hepatitis B Virus - Natural Killer
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHB patients (Other): a blood sample is done during a follow-up visit
  Interventions: Other: blood sample CHB patients
- Control group (Other): a blood sample
  Interventions: Other: boold sample Control group

INTERVENTIONS:
Other: blood sample CHB patients — During a boold sample at only one follow up visit:
  * 3 tubes EDTA 10 ml per patient
  * 1 tube "Paxgene" 1ml
  * 1 dry tube per patient
  Arms: CHB patients
Other: boold sample Control group — * 2 tubes EDTA ideally age and sex matched to CHB patient.
  * 1 tube "Paxgene" 1ml
  * 1 dry tube
  Arms: Control group

SUMMARY:
Natural Killer (NK) cells play a large role in the innate immune response as they are equipped to kill infected or tumor cells. They express a panel of activating and inhibitory receptors that regulate the destruction of the target cell. Many reports have shown that NK cell function is suppressed in CHB patients. Exhaustion occurs when activating receptors become over stimulated leading to the loss of NK function. The investigators hypothesize that NK cells are rendered dysfunctional/ exhausted by HBV. The primary objective is to determined the phenotypical modifications and mechanisms associated to NK cell dysfunction, during different phases of CHB infection, in not treated patients.

DETAILED DESCRIPTION:
Using a previous cohort from the Limoges Hospital, the investigators have identified by multi-parametric flow cytometry phenotypic, cytokine and signaling molecules that are altered in NK cells from CHB patients during the inactive phase. Phenotypic changes observed include the downregulation of CD160, NKp30, CD16 and Tim-3. The expansion of 'adaptive' NK cells (FCεRg- NKG2C+ or CD57hi), and the upregulation of CD107a (steady state), NKG2D and 41BB. Functional changes include the decrease in the levels of IFNγ, TNFα and MIP1β. Cellular metabolism is now recognized to regulate functional properties of immune cells such as T or NK cells. The mammalian target of rapamycin (mTOR) kinase is a key regulator of cellular metabolism, integrating environmental cues to control downstream metabolic pathways. mTOR is the catalytic subunit of two different complexes: mTORC1 and mTORC2, the activity of which can be measured by measuring the level of phosphorylation of the proteins S6 and Akt respectively. The lab has previously shown that the mTOR pathway regulates NK cell development and activation 2. The investigators have observed that pS6 and pAkt are also decreased in CHB patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

* Male or female, age ≥18 years
* HBV infection or chronic HBV infection
* Willing and able to provide written informed consent

Healthy donors must meet all of the following inclusion criteria to be eligible for participation in this study:

* Male or female, age between 18 and 50 years
* Willing and able to provide written informed consent

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:
* Infection with hepatitis C virus (HCV) or human immunodeficiency virus (HIV)
* Chronic liver disease of a non-HBV etiology
* Immune or cancerous disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Using a multiparameter flow cytometry approach, we will assess the mean fluorescence intensity (MFI) of the listed molecules expressed on Natural Killer cells | At inclusion, day 0

CONTACTS AND LOCATIONS:
Overall Officials: Véronique LOUSTAUD-RATTI, MD, Principal Investigator — Limoges Hospital; Uzma HASAN, Study Director — Inserm U1111, Lyon
Locations (1):
- Limoges Hospital, Limoges, France